CLINICAL TRIAL: NCT03115983
Title: A Concurrently Controlled Study of the LimiFlex™ Paraspinous Tension Band in the Treatment of Lumbar Degenerative Spondylolisthesis With Spinal Stenosis
Brief Title: LimiFlex Clinical Trial for the Treatment of Degenerative Spondylolisthesis With Spinal Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Empirical Spine, Inc. (Industry)
Collaborators: Biomedical Statistical Consulting (Unknown); Medical Metrics Diagnostics, Inc (Industry); MCRA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSS17001
Record Dates: First submitted 2017-03-31; First posted 2017-04-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Degenerative Spondylolisthesis; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Decompression; Gene Fusion

STUDY DESIGN:
Intervention Model Description: This is a multi-center, prospective, concurrently controlled, non-blinded study. Balance between groups will be achieved through sub classification using propensity scores. Prospective patient sample supplemented with retrospective and/or historical control subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LimiFlex (Experimental): Posterior dynamic stabilization with the LimiFlex Paraspinous Tension Band
  Interventions: Device: LimiFlex; Procedure: Decompression
- Fusion (Active Comparator): Transforaminal lumbar interbody fusion with concomitant posterolateral fusion with pedicle screw instrumentation
  Interventions: Device: Fusion Instrumentation; Procedure: Decompression; Procedure: Fusion

INTERVENTIONS:
Device: LimiFlex — LimiFlex implantation at a single level after surgical decompression.
  Other Names: LimiFlex Paraspinous Tension Band
  Arms: LimiFlex
Device: Fusion Instrumentation — Titanium alloy top-loading, polyaxial pedicle screws and cylindrical, titanium alloy rod instrumentation using autograft and/or allograft bone (i.e., cancellous and/or corticocancellous bone only), and/or a synthetic bone graft extender that is on-label for these indications (i.e., decorticated posterolateral gutter only). The TLIF requires a single PEEK or Titanium TLIF cage cleared by FDA for this indication filled with autograft and/or allograft bone (i.e., cancellous and/or corticocancellous bone only).
  Arms: Fusion
Procedure: Decompression — Surgical decompression at one or two contiguous levels from L1 to S1.
Procedure: Fusion — Transforaminal lumbar interbody fusion (TLIF) with concomitant posterolateral fusion (PLF) at a single level after surgical decompression.
  Arms: Fusion

SUMMARY:
The LimiFlex™ Clinical Trial is a prospective, concurrently controlled, multi-center study to evaluate the safety and effectiveness of decompression and stabilization with the Empirical Spine LimiFlex™ Paraspinous Tension Band compared to decompression and transforaminal lumbar interbody fusion (TLIF) with concomitant posterolateral fusion (PLF) for the treatment of lumbar degenerative spondylolisthesis (Grade I per Meyerding classification) with spinal stenosis. Clinical trial sites will enroll solely LimiFlex subjects or solely TLIF/PLF subjects.

DETAILED DESCRIPTION:
The LimiFlex™ Paraspinous Tension Band is a new stabilization option for patients being treated with surgical decompression for degenerative spondylolisthesis. The LimiFlex does not require pedicle screws to anchor to the spine; instead, two dynamic rods are attached to pedicle-sparing straps which encircle adjacent spinous processes.

ELIGIBILITY:
Inclusion Criteria (patients must meet ALL of the following criteria to be eligible for participation in the study):

1. Lumbar degenerative spondylolisthesis (Grade I per Meyerding classification), at one level from L1 to S1, with radiographic confirmation using X-ray;

   a. Grade I spondylolisthesis per Meyerding classification includes up to 25% anterior translation of a vertebra relative to the superior endplate of the subjacent vertebra at the index level. A patient is considered to have spondylolisthesis with a minimum 10% anterolisthesis at the affected level in a lateral x-ray image.
2. Lumbar spinal stenosis requiring decompression at up to two contiguous levels from L1 to S1, inclusive of the level diagnosed with degenerative spondylolisthesis, and confirmed radiographically using CT or MRI;

   a. At the index level, lumbar spinal stenosis is at least moderate lumbar canal stenosis, defined as more than 25% reduction of the cross-sectional area compared with the next adjacent normal level, with nerve root crowding compared with the normal level, as determined by the investigator on CT Scan or MRI.
3. Neurogenic claudication or radiculopathy symptoms including leg pain, muscle weakness, and/or sensation abnormality, with or without back pain as evidenced by patient history;
4. Persistent symptoms despite at least 3 months of conservative treatment that may include but is not limited to physical therapy, medications, and/or epidural injections;
5. A pre-operative Visual Analog Scale (VAS) leg pain score of ≥50 on a 100 mm scale;

   * Leg pain includes hip and/or buttock pain on the same side
6. A pre-operative Oswestry Disability Index (ODI) score ≥35 points on a 100-point scale;
7. Candidate for surgical decompression at a single level or two contiguous levels, with stabilization at only one level between L1-S1;
8. Posterior element anatomy is appropriate for interspinous fixation including prediction of presence of spinous processes of segment to be instrumented following decompression (investigational AND control groups) and a prediction of >50% of facet joints present following decompression (investigational group only);
9. ≥25-80 years of age and skeletally mature;
10. Patient has the necessary mental capacity to participate and is willing and able to participate in the study for the duration of the study follow-up and is able to comply with study requirements; and
11. Patient is willing to provide Informed Consent for study participation.

Exclusion Criteria:

1. A primary and predominate diagnosis of discogenic back pain;
2. A primary and predominate diagnosis of facet-mediated back pain;
3. Back or non-radicular leg pain of unknown etiology;
4. Significant peripheral vascular disease causing vascular claudication;
5. Significant peripheral neuropathy caused by conditions other than spinal stenosis;
6. History of fixed or permanent neurological deficit related to spinal cord injury;
7. History of any previous surgery* at any level in the lumbosacral spine except for a discectomy or decompression;
8. History of any previous surgery* at the level planned for treatment;

   * previous surgery includes spinal stimulator placement but does NOT include epidural injections, rhizotomy or nerve ablation.
9. Isthmic spondylolisthesis or spondylolysis (pars fracture) at any level in the lumbar spine;
10. Clinically significant compromise of vertebrae at L1 to S1 levels due to osteoporotic vertebral compression fracture or any traumatic, neoplastic, metabolic or infectious pathology or congenital abnormality;
11. Spinous process fracture(s) or other posterior element fracture(s) of the segment to be instrumented that would preclude secure fixation of the LimiFlex Device to the spinous process;
12. Spinous process insufficiency or deformity that would preclude secure fixation of the LimiFlex Device to the spinous process including spinous process length <10 mm from lamina to dorsal tip or other significant deformity due to trauma, or congenital abnormality such as spina bifida occulta at the planned instrumented level that would preclude secure fixation of the LimiFlex Device to the spinous process;
13. The estimated distance between the LimiFlex Device strap attachment points (midpoint of the cranial edge of the cranial spinous process and the midpoint of the caudal edge of the caudal spinous process) is <30mm on pre-operative lateral standing radiographs at the segment to be instrumented;
14. Degenerative lumbar scoliosis with a Cobb angle >10° at the affected motion segment;
15. Symptomatic lumbar stenosis that is not amenable to a direct decompression
16. Anklyosed motion segment at the target operative level
17. Severe osteoporosis, defined as history of fragility fracture and DXA T-score <-2.5 or QCT T-score <80mg/cubic cm. History of a fragility fracture requires that a DXA scan or QCT scan is completed;
18. Planned hip or knee replacement surgery, severe osteoarthritis or other musculoskeletal pathology of the hip or leg that could preclude reliable patient self reporting assessment scales and/or that would likely progress to surgery during study period;
19. Documented allergy to titanium or polyethylene;
20. Active local or systemic infection;
21. Receiving immunosuppressive or long-term steroid therapy;
22. Known history of bone metabolic disorder, including Paget's disease, hyperparathyroidism, renal osteodystrophy, and osteomalacia;
23. Disease or condition that would preclude accurate clinical evaluation of the safety and effectiveness of the study treatment or any significant medical conditions which would place the patient at excessive risk for surgery, such as:

    1. severe rheumatoid arthritis or other severe autoimmune disease
    2. active hepatitis (viral or serum) or HIV positive
    3. unstable cardiac disease
    4. uncontrolled diabetes
    5. renal failure
    6. severe muscular, neural or vascular diseases that endanger the spinal column
    7. cauda equina syndrome
    8. severe neurologic disorders including paralysis
24. Morbid obesity defined as BMI >40;
25. Active malignancy or history of metastatic malignancy within the last five years;
26. Women who are pregnant or are interested in becoming pregnant within the study period;
27. Currently seeking or receiving worker's compensation for back pain or spinal condition;
28. Currently involved in spinal litigation that potentially is associated with secondary financial gain;
29. Current involvement in a study of another investigational product for similar purpose;
30. Demonstrates three or more Waddell's Signs of Inorganic Behavior;
31. Active treatment of a major psychiatric condition, such as major depression, anxiety disorder, bipolar disorder, schizophrenia, personality disorder, that could prevent accurate completion of self reporting assessment scales;
32. Current history (within 12 months) of substance abuse, including alcohol abuse; or
33. A prisoner.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Success | 24 Months
  Individual success for patients in the investigational LimiFlex or control fusion arm is assessed with Composite Clinical Success (CCS) criteria. To be considered a success, a subject must demonstrate all of the following:
  * 15 point improvement in Oswestry Disability Index (100 point scale)
  * Absence of a new or worsening, persistent neurological deficit
  * Absence of additional surgical intervention
  * Absence of device integrity failures

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Oswestry Disability Index (ODI)
Neurological Status | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Neurological Status
Additional surgical interventions | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Additional surgical interventions
Absence of device integrity failures defined as device breakage, device separation or disassembly, or device dislocation | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Absence of device integrity failures defined as device breakage, device separation or disassembly, or device dislocation
Estimated blood loss | Procedure
  estimated blood loss and units of blood transfused
Length of procedure | Procedure
  Length of procedure (skin to skin)
Hospital stay | Immediately upon discharge
  Hospital stay
Return to normal activities of daily living | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Length of time for subject to return to his/her normal activities of daily living.
Work status | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Work status and days to return to work (as appropriate)
Pain medication including narcotics usage | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Medication use for pain, including narcotic, usage
Visual analog scale (VAS) leg pain | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Leg pain as measured on a Visual Analog Scale (VAS)
Visual analog scale (VAS) back pain | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Back pain as measured on a Visual Analog Scale (VAS)
Zurich claudication questionnaire (ZCQ) | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Zurich claudication questionnaire
SF-12 Quality of Life survey | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  SF-12 Health Survey
Patient satisfaction | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Patient satisfaction questionnaire
Radiographic fusion status | Both groups: 6 wks, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo, 48 mo, 60 mo
  Radiographic fusion status

CONTACTS AND LOCATIONS:
Overall Officials: Rick Sasso, MD, Principal Investigator — Indiana Spine Group; William C Welch, MD, Principal Investigator — Pennsylvania Hospital Neurosurgery
Locations (28):
- United States (28):
  - Sonoran Spine Research and Education Foundation, Tempe, Arizona
  - Kaiser Permanente Division of Research, Oakland, California
  - Stanford University Medical Center, Redwood City, California
  - UC Davis Spine Center, Sacramento, California
  - Kaiser Permanente Roseville Clinical Trials Program, Sacramento, California
  - UCSF Dept of Orthopaedic Surgery, San Francisco, California
  - Kaiser Permanente (San Jose Medical Center), San Jose, California
  - The Spine Institute, Center for Spinal Restoration and Foundation for Spinal Restoration, Santa Monica, California
  - Boulder Neurological & Spine Associates, Boulder, Colorado
  - University of Miami, Dept of Neurological Surgery, Miami, Florida
  - BioSpine, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Dept of Orthopedics and Physical Rehabilitation, Worcester, Massachusetts
  - Beaumont Hospital, Royal Oak, Michigan
  - Michigan Minimally Invasive Neurosurgical Institute, Waterford, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - UHS Neurosurgery (Binghamton), Binghamton, New York
  - Hospital for Special Surgery, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Texas Back Institue, Clincal Research, LLC-Plano, Plano, Texas
  - University of Virginia Orthopaedic Surgery, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maislin G, Keenan BT, Alamin TF, Fielding LC, Scherman A, Hachadoorian R, Pierre C, Sasso RC, Lavelle WF, Chapman J. Are Randomized Trials Better? Comparison of Baseline Covariate Balance of a Propensity Score-Balanced Lumbar Spine IDE Trial and Comparable RCTs. Global Spine J. 2025 Jul;15(6):2923-2930. doi: 10.1177/21925682251316287. Epub 2025 Jan 27. PMID 39868633